CLINICAL TRIAL: NCT00061451
Title: ALIMTA Plus Gemcitabine as Front-line Chemotherapy for Patients With Locally Advanced or Metastatic Non-Small-Cell Lung Cancer: A Phase II Clinical Trial
Brief Title: Pemetrexed Plus Gemcitabine as Front-Line Chemotherapy for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7213; H3E-US-JMFY
Record Dates: First submitted 2003-05-28; First posted 2003-05-29 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Gemcitabine

INTERVENTIONS:
Drug: Pemetrexed
Drug: Gemcitabine

SUMMARY:
The purposes of this study are to determine:

1. The safety of Pemetrexed plus Gemcitabine and any side effects that might be associated with the combination of these two drugs.
2. Whether Pemetrexed plus Gemcitabine can help patients with non-small cell lung cancer live longer.
3. Whether Pemetrexed plus Gemcitabine can make the tumor smaller or disappear, and for how long.
4. To see if patients feel better while taking Pemetrexed plus Gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Non-Small Cell Lung Cancer that can be treated with chemotherapy.
* Have received no prior chemotherapy for Non-Small Cell Lung Cancer.
* Have at least one measurable lesion.
* Have an adequate performance status.
* Sign an informed consent.

Exclusion Criteria:

* A female who is pregnant or breastfeeding.
* Treatment with an investigational drug within the last 30 days, previously completed or withdrawn from this study or any other study investigating Pemetrexed.
* Treatment with radiation therapy within the last 4 weeks.
* Brain metastasis that is uncontrolled.
* Active infection or other serious condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2002-12; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To assess the objective tumor response rate of gemcitabine plus pemetrexed in patients with advanced or metastatic non-small-cell lung cancer.

SECONDARY OUTCOMES:
To assess time to objective tumor response for responding patients
To assess duration of response for responding patients
To assess time to treatment failure for patients
To assess progression free survival of patients
To assess time to progressive disease for patients
To assess survival time for patients
To characterize the toxicities of gemcitabine plus pemetrexed in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Falls, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559 or 317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com